CLINICAL TRIAL: NCT06112249
Title: Efficacy of the SAFE Program to Promote Preventative Behaviors of Airborne Diseases (COVID-19) and Improve Well-Being for People With Intellectual and Developmental Disabilities in the Workplace
Brief Title: SAFE Workplace Intervention for People With IDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 27789
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Communicable Diseases; Prevention; Workplace Intervention
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Three arm study with a control group, a peer interventionist group and staff delivered group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The statistician will blindly randomize the three arm groups. The only staff with access to the groups will be the research coordinator. The primary investigators are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Does not receive curriculum.
- Peer Intervention (Experimental): Receives curriculum taught by Peer Interventionist
  Interventions: Behavioral: SAFE Employment Training
- Staff Delivered (Experimental): Receives curriculum taught by staff
  Interventions: Behavioral: SAFE Employment Training

INTERVENTIONS:
Behavioral: SAFE Employment Training — The SAFE program includes lessons in the following areas: 1) Overview of What COVID-19 is and how it spreads 2) What is PPE and How to properly use 3) Social Distancing 4) Community Participation 5) Employment 6) Self Efficacy. We would also like to know if you learn more when the SAFE program is taught by a peer (person who also has an intellectual developmental disability).
  Arms: Peer Intervention; Staff Delivered

SUMMARY:
The purpose of this study is to examine the feasibility and efficacy of a systematic training approach targeting behaviors to increase safety and prevention of airborne diseases such as COVID-19 in the workplace for individuals with Intellectual and Developmental Disabilities (IDD). This project is designed to determine proof of concept and proof of product for a peer support intervention, the SAFE program, to increase knowledge and safe workplace practices. There is an identified immediate need for individuals with IDD to receive training in an accessible format. The SAFE program has been developed in an accessible format for those with IDD. It focuses on education regarding actionable behaviors that reduce the risk of acquiring and transmitting COVID-19 and other airborne diseases. The study will implement a peer-mediated and occupational therapy lead program, SAFE, to identify and address potential implementation issues and further refine the program curriculum. Additionally, the efficacy of the program on perceived safety and well-being, observable preventative behaviors and self-advocacy will be examined.

DETAILED DESCRIPTION:
It is hypothesized that the SAFE program will have a positive effect on perceived well-being and knowledge of the actionable behaviors for the prevention of COVID-19 and other airborne diseases. The program will have a larger effect on outcomes when provided using peer support compared to staff training. Individuals with IDD will demonstrate increased knowledge and safe behaviors after completing the SAFE program. Peer-interventionists will report perceived benefits and limitations of participating in training and providing peer-mediated travel training interventions to identify potential outcomes for future research.

The research intends to answer these questions:

Does participation in the SAFE program increase perceived safety and well-being in the workplace for people with Autism Spectrum Disorder (ASD) and/or Intellectual or Developmental Disabilities (IDD)? Does participation in the SAFE program increase knowledge of actionable behaviors to prevent transmission of airborne diseases (i.e. COVID-19) in the workplace for people with IDD? When implemented through peer support, does the SAFE program have a larger increase in perceived well-being and knowledge of actionable behaviors to prevent transmission of airborne diseases (i.e. COVID-19) than when implemented through staff training and supports?

The research further intends to:

Develop health communication messages related to safe interactions and the prevention of COVID-19 and other infectious airborne diseases for autistic adults

Refine and expand the SAFE program based on stakeholder priorities and input

Evaluate the SAFE program training with Autistic adults Procedures.

The researchers will leverage current relationships with community organizations to recruit 100 participants with ASD and or IDD who are employed 10 hours or more a week and receiving employment services or supports. Organizational administrators will provide information on the study to individuals that meet the inclusion criteria. Interested individuals will contact the project research coordinator to determine inclusion. Eligible participants will be randomized into one of the 3 arms of the study, Control, Peer Interventionist Led, Staff Led.

If the participant is assigned to the staff intervention support staff will be contacted with an email or phone call. Staff members will be required to complete human subjects training. Researchers will obtain informed consent for all participants. During the first contact made with participants, written information will be provided remotely using Zoom/FaceTime or in person to all participants explaining the following in simple terms: 1) the criteria for participation, 2) the purpose of the research and the procedures involved, 3) the subject's right to withdraw at any time without penalty of any sort, 4) potential benefits to the subject, 5) potential risks, 6) assurance of anonymity, and 7) terms of remuneration. All research staff will complete training about the informed consent process prior to consenting subjects. The information described above will be reviewed and any questions answered. Participants will be obtained signed or a printed signature box used for signature when electronic signatures are unable to be obtained for consent either in person or virtually.

The researchers will collect data from young adults or transitional aged-youth with ASD or IDD to determine the efficacy and feasibility of the intervention. Recruitment occurs through the sites identified in the participant recruitment section of this proposal. Participants interested in the study will contact the primary investigator or research staff who will schedule an initial physical or virtual meeting at a place and time convenient for the participant to determine inclusion and obtain consent/assent. Participants are randomly assigned to either peer-support intervention, staff intervention or a control group. The researchers will randomize in blocks of 12 (4 to each group) until the investigators reach the targeted number of 120 or 40 participants in each group. Pre-test and post-test measures will be administered by researcher staff prior to the start of the intervention (Pre-test) and at the end of the intervention 4 weeks (Post-test ). Key stakeholders, including the participants and interventionists (occupational therapists and peer mediators), will complete qualitative interviews at the end of the intervention period for each participant. The information gathered will determine acceptability and feasibility of intervention. Participants will be asked to discuss their experiences during the intervention specific to their assigned intervention group.

A member from the research team will then contact interested individuals to set up a convenient meeting time and place for the SAFE program training. These meetings will occur remotely or in a private location convenient to the participant. The SAFE program course training will occur in small group settings or individually. The course trainings will occur 2-3 times per week for between 45-60 minutes. An appropriate curriculum has been developed by Temple University Researchers and Occupational therapy students based on many qualitative interviews, research of proper education methods, and COVID-19 practices. The curriculum is based on a series of classes designed to create an understanding of best practices and behaviors to prevent the spread of COVID-19 in the workplace. The curriculum will be adapted to meet the needs of this project and study population. The course will provides instruction in the following areas: 1) COVID-19 and how it spreads 2) Personal Protective Equipment (PPE) and How to use it properly 3) Social Distancing 4) Community Participation 5) Employment 6) Self Efficacy.

Participants will complete the SAFE program sessions remotely or in person in a private, quiet and convenient setting.. Participants will be randomized into two treatment arms and a control group. The first treatment arm will receive the SAFE program implemented through a staff training model. The second group will receive the program using a peer support model. The control group will continue to receive their standard vocational rehabilitation supports.

Training of the SAFE program will occur remotely or in person by staff who are trained within our research team or will be implement it in collaboration with staff or a peer specialist remotely as part of their current services. If it is in person it will be implemented at their vocational rehabilitation centers or places of employment. Research staff will be available to support the process after the training is complete.

The researchers will use a questionnaire to assess knowledge of actionable behaviors to prevent COVID-19, which reflect the core components of the SAFE program (social distancing, proper use of PPE, personal hygiene practices, and self-advocacy in the workplace). The researchers will also administer measures to determine the degree of self-advocacy and self-efficacy in the work place reported by staff and self-reported by participants. The researchers will determine how well a participant follows workplace procedures. Data will be collected either in person or virtually both at pre-test and post-test for all outcome measures. Finally, the investigators will assess perceived anxiety.

ELIGIBILITY:
Inclusion Criteria:

* The researchers anticipate recruiting young adults 18years old and over with ASD or IDD who are currently employed or actively looking for employment to participate in the study. Participants will have a diagnosis of ASD or IDD. Participants will self-report their ASD or IDD diagnosis. Additionally, the community agencies have access to documentation that identifies their consumer's diagnoses. Based on this, the researchers will ask them to only provide information to those individuals who have a diagnosis of IDD. Potentially eligible participants with documented intellectual and developmental disabilities will be recruited through large vocational rehabilitation organizations (Community Integrated Services CIS and Project Search) that together serve over 1200 adults with IDD. Participants must be working a minimum of 10 hours a week outside the home and/or receive vocational rehabilitation services.

Exclusion Criteria:

* under 18 years, do not have a minimum of 10 hours/week of work experience, do not have Autism Spectrum Disorder and/or Intellectual Disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2025-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Pfeiffer, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - JEVS, Collingswood, New Jersey
  - Community Integrated Services, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfeiffer, B., Davidson, A., Kelly, P. J., Luck, C., Singley, K., & Bass, S. (2024). Infectious Airborne Disease Knowledge, Training Preferences, and Peer Support Acceptance among Young Working Autistic Adults: A Qualitative Inquiry. Journal of Vocational Rehabilitation, 10522263251337562.
- See also: A summary of the research study and links to SAFE Curriculum for Students and the SAFE Curriculum for Instructors. — https://sites.temple.edu/reachlabtemple/safe-social-distancing-and-advocacy-for-personal-protective-equipment-and-employment/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 67 participants were recruited from 10 agencies that provide services to young adults with intellectual and developmental disabilities in and around the Philadelphia area. Recruitment and enrollment took place from 10/2023 thru 2/2024.
Pre-assignment Details: No pre-assignment issues were encountered.
Groups:
- Control Group: Does not receive SAFE Curriculum
- Peer Intervention: Receives SAFE Curriculum taught by Peer Interventionist
- Staff Delivered: Receives SAFE Curriculum taught by staff.
Period: Overall Study
Arm/Group | Control Group | Peer Intervention | Staff Delivered
Started | 20 | 22 | 25
Completed | 20 | 22 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Peer Intervention | Staff Delivered | Total
Number analyzed (Participants) | 20 | 22 | 25 | 67
Age, Customized [Count of Participants; unit: Participants]
  18 - 20 years | 18 | 19 | 13 | 50
  21 - 26 years | 2 | 2 | 3 | 7
  27 - 38 years | 0 | 0 | 9 | 9
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3 | 4 | 0 | 7
  Male | 17 | 18 | 20 | 55
  Other | 0 | 0 | 4 | 4
  Missing Response | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5 | 10
  Not Hispanic or Latino | 17 | 20 | 20 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian and Pacific Islander | 5 | 2 | 3 | 10
  Native American/Alaska Native | 1 | 2 | 2 | 5
  Black/African American | 4 | 7 | 4 | 15
  White/Caucasian | 6 | 4 | 14 | 24
  Multiple Races | 1 | 3 | 0 | 4
  Other | 0 | 1 | 2 | 3
  Decline to answer | 2 | 1 | 0 | 3
  Missing Response | 1 | 2 | 0 | 3
Primary Disability [Count of Participants; unit: Participants]
  Intellectual Disability (ID) | 5 | 2 | 3 | 10
  Autism Spectrum Disorder (ASD) | 14 | 19 | 18 | 51
  Other Diagnosis | 0 | 0 | 2 | 2
  Decline to answer | 1 | 1 | 1 | 3
  Missing Response | 0 | 0 | 1 | 1
Highest Level of Education Completed [Count of Participants; unit: Participants]
  Completed up to grade 11 | 8 | 3 | 6 | 17
  High School Graduate or GED | 10 | 18 | 11 | 39
  Some college, vocational, trade or business School | 1 | 1 | 3 | 5
  Associates degree or vocational graduate | 0 | 0 | 1 | 1
  Bachelors degree | 0 | 0 | 2 | 2
  Some graduate of professional school training | 1 | 0 | 1 | 2
  Graduate or professional degree | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Infectious Airborne Disease Knowledge and Preventative Behaviors Outcomes
Description: The Infectious Airborne Disease Knowledge and Prevention of Behavior Outcomes is an assessment to see the knowledge of infectious airborne disease preventative behaviors gained through the SAFE curriculum. The assessment is completed through true and false questions, multiple choice questions, open ended questions, and behavior observations. Score: 1 - 67. Higher scores mean better outcomes.
Time Frame: Pre Data (before intervention), Post1 (immediately following), Post2 (1 month after)
Population: Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered").
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Peer Intervention | Staff Delivered
Number analyzed (Participants) | 20 | 22 | 25
score on a scale
  Pre Data (before intervention) | .61 (.17) | .71 (.15) | .72 (.12)
  Post 1 (immediately following): number analyzed (Participants) | 20 | 22 | 24
  Post 1 (immediately following) | .65 (.16) | .74 (.11) | .84 (.07)
  Post 2 (1 month after): number analyzed (Participants) | 20 | 20 | 24
  Post 2 (1 month after) | .66 (.17) | .75 (.13) | .83 (.06)
  Change from "Pre Data" at "Post 1": number analyzed (Participants) | 20 | 22 | 24
  Change from "Pre Data" at "Post 1" | 0.11 (0.12) | 0.04 (0.22) | 0.03 (0.12)
  Change from "Pre Data" at "Post 2": number analyzed (Participants) | 20 | 20 | 24
  Change from "Pre Data" at "Post 2" | 0.11 (0.12) | 0.04 (0.22) | 0.03 (0.12)
Statistical Analysis 1: Comparison: Control Group vs Peer Intervention vs Staff Delivered; One-Way ANCOVA mixed effect model is performed to compare the change score from "Pre Data" at "Post 1" among three groups. Linear mixed-effect model is used to compute test statistics and the overall significance. In each model, classroom (cluster-level) is included as random effects, and both age and education level are included as fixed covariates,; Test type: Superiority; p = 0.3094, Mixed Models Analysis — The threshold for statistical significance was p=0.05; A F-statistics=1.20 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education
Statistical Analysis 2: Comparison: Control Group vs Peer Intervention vs Staff Delivered; One-Way ANCOVA mixed effect model is performed to compare the change score from "Pre Data" at "Post 2" among three groups. Linear mixed-effect model is used to compute test statistics and the overall significance. In each model, classroom (cluster-level) is included as random effects, and both age and education level are included as fixed covariates,; Test type: Superiority; p = 0.3966, Mixed Models Analysis — The threshold for statistical significance was p=0.05; A F-statistics=0.94 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education

2. Secondary Outcome: Workplace Health and Safety Assessment
Description: This measure was adapted from employment-centered items on the Self-Determination and Self-Advocacy Questionnaire, which assess the degree of self-advocacy in the workplace as reported by staff and self-reported by participants. Score: 1 - 25. Higher scores mean better outcomes.
Time Frame: Pre Data (before intervention), Post1 (immediately following), Post2 (1 month after)
Population: Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered").
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Peer Intervention | Staff Delivered
Number analyzed (Participants) | 20 | 22 | 25
score on a scale
  Pre Data (before intervention): number analyzed (Participants) | 20 | 21 | 25
  Pre Data (before intervention) | 3.68 (1.08) | 2.99 (1.14) | 3.74 (.84)
  Post 1 (immediately following): number analyzed (Participants) | 20 | 22 | 24
  Post 1 (immediately following) | 3.43 (1.19) | 3.43 (1.04) | 3.84 (.82)
  Post 2 (1 month after): number analyzed (Participants) | 20 | 20 | 23
  Post 2 (1 month after) | 3.35 (1.26) | 3.72 (.95) | 4.03 (.70)
  Change from "Pre Data" at "Post 1": number analyzed (Participants) | 20 | 21 | 24
  Change from "Pre Data" at "Post 1" | -0.25 (0.79) | 0.45 (1.10) | 0.10 (0.74)
  Change from "Pre Data" to "Post 2": number analyzed (Participants) | 20 | 19 | 23
  Change from "Pre Data" to "Post 2" | -0.15 (0.82) | 0.79 (1.21) | 0.31 (0.76)
Statistical Analysis 1: Comparison: Control Group vs Peer Intervention vs Staff Delivered; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0491, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=3.20 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education
Statistical Analysis 2: Comparison: Control Group vs Peer Intervention vs Staff Delivered; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0264, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=3.93 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) General Self-Efficacy Item Bank
Description: This measure assesses a person's belief in their capacity to manage daily stressors and have control over meaningful events. Participants will complete the 10-question tool which is designed for people 18 years and older. It has established acceptable reliability and validity.81 The responses are on a 5 point scale from "never" (1) to "very often" (5) with higher scores reflecting greater general self-efficacy. The scale (average across 10 questions) ranges from 1 to 5.
Time Frame: Pre Data (before intervention), Post1 (immediately following), Post2 (1 month after)
Population: Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered").
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Peer Intervention | Staff Delivered
Number analyzed (Participants) | 20 | 22 | 25
score on a scale
  Pre Data (before intervention): number analyzed (Participants) | 20 | 20 | 25
  Pre Data (before intervention) | 3.20 (.94) | 3.30 (.90) | 3.38 (.75)
  Post 1 (immediately following): number analyzed (Participants) | 20 | 22 | 24
  Post 1 (immediately following) | 3.26 (1.03) | 3.21 (.85) | 3.39 (.77)
  Post 2 (1 month after): number analyzed (Participants) | 20 | 20 | 24
  Post 2 (1 month after) | 2.13 (1.12) | 3.31 (.77) | 3.25 (.78)
  Change from "Pre Data" at "Post 1": number analyzed (Participants) | 20 | 20 | 24
  Change from "Pre Data" at "Post 1" | 0.06 (0.56) | -0.07 (0.42) | 0.01 (0.45)
  Change from "Pre Data" to "Post 2": number analyzed (Participants) | 20 | 18 | 24
  Change from "Pre Data" to "Post 2" | -0.07 (0.89) | 0.03 (0.58) | -0.13 (0.72)
Statistical Analysis 1: Comparison: Control Group vs Peer Intervention vs Staff Delivered; Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered"); Test type: Superiority — One-Way ANCOVA mixed effect model is performed to compare the change score from "Pre Data" at "Post 1" among three groups. Linear mixed-effect model is used to compute test statistics and the overall significance. In each model, classroom (cluster-level) is included as random effects, and both age and education level are included as fixed covariates,; p = 0.8026, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=0.22 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education
Statistical Analysis 2: Comparison: Control Group vs Peer Intervention vs Staff Delivered; Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered"); Test type: Superiority — One-Way ANCOVA mixed effect model is performed to compare the change score from "Pre Data" at "Post 2" among three groups. Linear mixed-effect model is used to compute test statistics and the overall significance. In each model, classroom (cluster-level) is included as random effects, and both age and education level are included as fixed covariates,; p = 0.9615, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=0.04 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education

4. Secondary Outcome: Vocational Fit Assessment Safety Subscale
Description: The Vocfit is an assessment tool used to measure the best fit for a worker with a job. The tool was specifically developed for individuals with developmental disabilities and has strong psychometric properties for this population. Participants will complete the 10-question tool which is designed for people 18 years and older. The responses are on a 3 point scale from "Low = you can do it but you need someone else to help you the whole time" (0) to "High = you can do it by yourself" (2) with higher scores reflecting better fit for a worker with a job. The scale (average across 10 questions) ranges from 0 to 2.
Time Frame: Pre Data (before intervention), Post1 (immediately following), Post2 (1 month after)
Population: Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered").
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Peer Intervention | Staff Delivered
Number analyzed (Participants) | 20 | 22 | 25
score on a scale
  Pre Data (before intervention): number analyzed (Participants) | 17 | 20 | 23
  Pre Data (before intervention) | 1.00 (.5) | 1.06 (.45) | 1.21 (.36)
  Post 1 (immediately following): number analyzed (Participants) | 20 | 22 | 24
  Post 1 (immediately following) | .90 (.52) | 1.12 (.42) | 1.05 (.44)
  Post 2 (1 month after): number analyzed (Participants) | 20 | 20 | 25
  Post 2 (1 month after) | 1.04 (.49) | 1.20 (.45) | 1.21 (.44)
  Change from "Pre Data" at "Post 1": number analyzed (Participants) | 17 | 20 | 22
  Change from "Pre Data" at "Post 1" | -0.12 (0.39) | 0.06 (0.43) | -0.19 (0.45)
  Change from "Pre Data" to "Post 2": number analyzed (Participants) | 17 | 18 | 22
  Change from "Pre Data" to "Post 2" | 0.05 (0.60) | 0.18 (0.35) | -0.03 (0.35)
Statistical Analysis 1: Comparison: Control Group vs Peer Intervention vs Staff Delivered; Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered"); Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.2128, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=1.60 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education
Statistical Analysis 2: Comparison: Control Group vs Peer Intervention vs Staff Delivered; Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered"); Test type: Superiority — [test comment as in outcome 3, analysis 2]; p = 0.4228, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=0.88 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education

5. Secondary Outcome: National Institutes of Health (NIH) Toolbox Item Bank/Fixed Form v2.0 - Perceived Stress (Ages 18+).
Description: This measure assesses "perceptions about the nature of events and their relationship to the values and perceived coping resources of an individual" for adults 18 years and older. This self-report measure has 10 items with a response range from "Never" (1) to "Very Often" (5). Higher scores reflect greater levels of perceived stress. The scale (average across 10 questions) ranges from 1 to 5.
Time Frame: Pre Data (before intervention), Post1 (immediately following), Post2 (1 month after)
Population: Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered").
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Peer Intervention | Staff Delivered
Number analyzed (Participants) | 20 | 22 | 25
score on a scale
  Pre Data (before intervention): number analyzed (Participants) | 20 | 21 | 25
  Pre Data (before intervention) | 2.87 (.37) | 2.98 (.41) | 3.11 (.54)
  Post 1 (immediately following): number analyzed (Participants) | 20 | 22 | 24
  Post 1 (immediately following) | 2.71 (.45) | 2.95 (.45) | 2.90 (.58)
  Post 2 (1 month after): number analyzed (Participants) | 20 | 20 | 25
  Post 2 (1 month after) | 2.66 (.45) | 2.93 (.49) | 3.04 (.59)
  Change from "Pre Data" at "Post 1": number analyzed (Participants) | 20 | 21 | 24
  Change from "Pre Data" at "Post 1" | -0.17 (0.53) | -0.01 (0.35) | -0.20 (0.47)
  Change from "Pre Data" to "Post 2": number analyzed (Participants) | 20 | 19 | 24
  Change from "Pre Data" to "Post 2" | -0.22 (0.50) | -0.04 (0.38) | -0.07 (0.44)
Statistical Analysis 1: Comparison: Control Group vs Peer Intervention vs Staff Delivered; Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered"); Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1943, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=1.69 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education
Statistical Analysis 2: Comparison: Control Group vs Peer Intervention vs Staff Delivered; Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered"); Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.3540, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=1.06 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 - Anxiety Short Form 8.
Description: This measure assesses anxiety for adults 18 years and older. This self-report measure has 8 items with a response range from "Never" (1) to "Always" (5). Higher scores reflect greater levels of anxiety. It has established acceptable psychometrics and is sensitive to change. The scale (average across 8 questions) ranges from 1 to 5.
Time Frame: Pre Data (before intervention), Post1 (immediately following), Post2 (1 month after)
Population: Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered").
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Peer Intervention | Staff Delivered
Number analyzed (Participants) | 20 | 22 | 25
score on a scale
  Pre Data (before intervention): number analyzed (Participants) | 20 | 21 | 25
  Pre Data (before intervention) | 18.25 (6.45) | 18.86 (7.51) | 20.82 (6.82)
  Post 1 (immediately following): number analyzed (Participants) | 20 | 22 | 24
  Post 1 (immediately following) | 20.15 (8.7) | 20.86 (6.77) | 20.79 (7.28)
  Post 2 (1 month after): number analyzed (Participants) | 20 | 20 | 24
  Post 2 (1 month after) | 17.25 (7.30) | 20.70 (7.49) | 21.21 (5.68)
  Change from "Pre Data" at "Post 1": number analyzed (Participants) | 20 | 21 | 24
  Change from "Pre Data" at "Post 1" | 1.90 (8.52) | 2.00 (6.22) | -0.13 (5.57)
  Change from "Pre Data" to "Post 2": number analyzed (Participants) | 20 | 19 | 24
  Change from "Pre Data" to "Post 2" | -1.00 (5.70) | 2.32 (9.85) | 0.29 (4.46)
Statistical Analysis 1: Comparison: Control Group vs Peer Intervention vs Staff Delivered; Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered"); Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1842, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=1.75 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education
Statistical Analysis 2: Comparison: Control Group vs Peer Intervention vs Staff Delivered; Intent to treat population (all participants assigned to "Control", "Peer Intervention", "Staff Delivered"); Test type: Superiority — [test comment as in outcome 3, analysis 2]; p = 0.6832, Mixed Models Analysis — The threshold for statistical significance was p=0.05; p-value indicates overall significance among three groups; A F-statistics=0.38 is obtained for testing overall significance among three groups using mixed effect model, adjusted by age and education

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Control Group | Peer Intervention | Staff Delivered
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 0/25

LIMITATIONS AND CAVEATS:
The sample is limited to the Philadelphia area, reducing generalizability. Randomization occurred by classroom, not individual, which may have influenced responses due to differences in support needs. One classroom had higher overall support, possibly affecting how lessons were accessed and surveys completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT06112249/Prot_SAP_000.pdf